CLINICAL TRIAL: NCT04706650
Title: Exercise Capacity in Axial Spondyloarthritis and Factors Affecting it: a Cross-sectional Controlled Study
Brief Title: Exercise Capacity, Cardiovascular Risk Factors and Disease-related Variables in Axial Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ebru Koseoglu Tohma, specialist medical doctor, Muğla Sıtkı Koçman University
Other Study IDs: muğla sıtkı koçman university
Record Dates: First submitted 2021-01-05; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Exercise Capacity; Axial Spondyloarthritis
Keywords: axial spondyloarthritis; exercise capacity; cardiovascular risk factors; nonradiographic axial spondyloarthritis; cardiorespiratory fitness
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to study the associations between exercise capacity and cardiovascular (CV) risk factors in axial spondyloarthritis (axSpA) patients and to determine possible relationships with disease-related variables. Thirty eight patients and 38 controls were recruited in our cross-sectional controlled study. Comprehensive systemic and musculoskeletal examinations were carried out in both of the groups. Cardiovascular risk profile data, ASDAS-CRP, 10-year CV event risk, physical activity levels (IPAQ) were recorded. A maximal treadmill exercise test by Bruce protocol was administered to all participants.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of axial SpA
* must be able to walk

Exclusion Criteria:

* established cardiac disease including structural heart diseases,
* uncontrolled hypertension,
* cardiac rhythm disorder,
* unstable angina pectoris,
* chronical renal and/or hepatic disease,
* malignancy,
* neuromuscular disease
* musculoskeletal deformity
* the history of an inflammatory arthritis for control group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty eight patients fulfilling the ASAS axial SpA criteria were recruited from the department of Gazi University Physical Medicine and Rehabilitation Rheumatology. 38 control subjects were randomly recruited from local hospital staff with a similar range of sex and age to the patients.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2014-10-15 (Actual)

PRIMARY OUTCOMES:
Mean difference in exercise capacity of axSpA patients and controls | may- october 2014
  maximal METs achieved by a maximal treadmill test by Bruce protocol

SECONDARY OUTCOMES:
Mean difference in heart rate recovery of axSpA patients and controls | may- october 2014
  peak heart rate achieved by maximal exercise minus heart rate at 1st minute of recovery phase